CLINICAL TRIAL: NCT07161037
Title: A Phase 2a, Open-label, Single-arm Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of VX-407 in Subjects With Autosomal Dominant Polycystic Kidney Disease Who Have a Subset of PKD1 Gene Variants
Brief Title: Phase 2a Study of VX-407 in Participants With ADPKD Who Have a Subset of PKD1 Gene Variants (AGLOW)
Acronym: AGLOW
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-407-101; 2024-517393-13-00 (Other: EU CTIS)
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX-407 (Experimental): Participants will receive VX-407 for up to 52 weeks.
  Interventions: Drug: VX-407

INTERVENTIONS:
Drug: VX-407 — Tablets for oral administration.

SUMMARY:
The purpose of the study is to evaluate the effect of VX-407 on height-adjusted total kidney volume (htTKV), safety, tolerability, and pharmacokinetics (PK) of VX-407.

ELIGIBILITY:
Key Inclusion Criteria:

* A pre-existing diagnosis of ADPKD as defined in the protocol
* Willing and able to comply with scheduled visits and other study procedures
* Participants with ADPKD with Mayo imaging classification (MIC) status of 1B (with htTKV ≥250 mL/m), 1C, 1D, or 1E confirmed by abdominal MRI obtained during screening
* Estimated glomerular filtration rate (eGFR) greater than or equal to (≥) 25 milliliter per minute (mL/min)/1.73 square meter (m^2)

Key Exclusion Criteria:

* History of kidney disease other than ADPKD that in the opinion of the investigator would independently impact the natural history of ADPKD
* History of solid organ or bone marrow transplantation or nephrectomy
* Ongoing renal replacement therapy or planning to start renal replacement therapy within 12 months of screening

Other protocol defined Inclusion/Exclusion criteria will apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
htTKV on MRI Over Time | Baseline up to End of Study (Week 52)

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Week 54
Maximum Observed Plasma Concentration (Cmax) of VX-407 | From Day 1 up to Week 52
Area Under the Concentration Versus Time Curve (AUC) of VX-407 | From Day 1 up to Week 52

CONTACTS AND LOCATIONS:
Locations (29):
- United States (20):
  - Alabama Kidney Research, Alabaster, Alabama
  - University of Alabama at Birmingham- Nephrology Research Clinic, Birmingham, Alabama
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCSF Clinical Research Center at Parnassus, San Francisco, California
  - Nephrology & Hypertension Associates, PC, Middlebury, Connecticut
  - Yale University - Yale Nephrology Clinical Research Clinic, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory School of Medicine - Renal Division, Atlanta, Georgia
  - Renal Associates, Columbus, Georgia
  - UChicago Medicine - Duchossois Center for Advanced Medicine - Nephrology, Chicago, Illinois
  - University of Iowa Health Care Medical Center- Nephrology, Iowa City, Iowa
  - The University of Kansas Medical Center Division of Nephrology, Kansas City, Kansas
  - University of Maryland Medical Center - General Clinical Research Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center - Nephrology, Boston, Massachusetts
  - University of Minnesota -Clinics and Surgery Center (CSC) - Endocrine Clinic, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - DaVita Kidney Care - Las Vegas, Las Vegas, Nevada
  - Columbia University Medical Center/NYP, New York, New York
  - UVM Medical Center - 1 South Prospect Street, Burlington, Vermont
- Belgium (2):
  - Universite Catholique de Louvain - Nephrology, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg - Nephrology, Leuven
- McGill University Health Centre, Montreal, Canada
- Centre Hospitalier Regional Universitaire (CHRU) Brest, Brest, France
- United Kingdom (5):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - King's College Hospital - Pulmonology, London
  - Royal Free Hospital - Nephrology, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital - Nephrology, Newcastle upon Tyne
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/